CLINICAL TRIAL: NCT06599307
Title: The Effect of Rituximab on Cognitive and Hand Functions in Secondary Progressive Multiple Sclerosis: a Randomized Controlled Trial
Brief Title: The Effect of Rituximab on Cognitive and Hand Functions in Secondary Progressive Multiple Sclerosis
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Amgad Mahmoud Elmeligy, Assistant lecturer of Neurology, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: MD-146-2024
Record Dates: First submitted 2024-09-10; First posted 2024-09-19 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Secondary Progressive Multiple Sclerosis (SPMS)
Keywords: Rituximab; Cognitive functions; Hand functions; Secondary Progressive Multiple Sclerosis
MeSH Terms: conditions — Multiple Sclerosis, Chronic Progressive | interventions — Rituximab; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intervention (Experimental): This group will receive Rituximab as follows: initial 1gm divided into 2 doses (500 mg each) given 2 weeks apart then another 1gm will be given after 6 months. Vials will be diluted on 500 ml normal saline 0.9% and will be given as intravenous infusions.
  Interventions: Drug: Rituximab
- Control (Placebo Comparator): This group will receive 500 ml normal saline 0.9% as intravenous infusions. Another dose will be given after 6 months
  Interventions: Other: Saline (NaCl 0,9 %) (placebo)

INTERVENTIONS:
Drug: Rituximab — Rituximab 1gm vial diluted on 500 ml normal saline 0.9%
  Arms: Intervention
Other: Saline (NaCl 0,9 %) (placebo) — 500 ml of normal saline 0.9%
  Arms: Control

SUMMARY:
The goal of this clinical trial is to know if rituximab can improve cognitive and hand functions in secondary progressive multiple sclerosis (SPMS) patients with high disability (EDSS 6.5 or more). The main questions it aims to answer are:

Can rituximab improve cognitive and hand functions in SPMS patients? Can rituximab improve the quality of life and the Expanded Disability Status Scale (EDSS) in SPMS patients?

Researchers will compare patients who receive rituximab to patient who receive placebo to see the effects of rituximab on cognition, hand functions, quality of life and EDSS.

Demographic and clinical data as age, gender, disease duration and EDSS will be obtained from each participant. Participants will perform The Brief International Cognitive Assessment for Multiple Sclerosis (BICAMS), The Nine-Hole Peg Test (9-HPT) and The MS-QLQ27 questionnaire at baseline and after one year of receiving either rituximab or placebo.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosis of secondary progressive multiple sclerosis by Lorscheider et al's criteria (disability progression by 1 EDSS step in patients with EDSS ≤ 5.5 or 0.5 EDSS step in patients with EDSS ≥ 6 in the absence of a relapse, a minimum EDSS score of 4 and pyramidal functional system (FS) score of 2 and confirmed progression over ≥3 months, including confirmation within the leading FS).
2. Baseline EDSS ≥ 6.5.

Exclusion Criteria:

1. Patients received disease modifying therapy for SPMS other than rituximab.
2. Clinical relapse in the last 3 months before recruitment.
3. Patients with documented hypersensitivity or contraindication to rituximab.
4. Patients with concomitant neurologic conditions that may affect cognitive or hand functions.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 46 (Estimated)
Dates: Start 2024-08-01 (Actual); Primary Completion 2026-05 (Estimated); Study Completion 2026-05 (Estimated)

PRIMARY OUTCOMES:
The effect of rituximab on cognitive functions assessed by The Symbol Digit Modalities Test | One year
  The Symbol Digit Modalities Test (SDMT) presents a series of nine symbols, each paired with a single digit in a key at the top of a standard sheet of paper. Patients are asked to identify the digit associated with each symbol as rapidly as possible for 90 seconds. The outcome measure is the number of correct responses over the 90 seconds time span.
The effect of rituximab on cognitive functions assessed by The Brief Visuospatial Memory Test-Revised | One year
  The Brief Visuospatial Memory Test-Revised (BVMT-R) constitutes of six abstract designs presented to the patient for 10 seconds. The display is removed from view and patients render the stimuli via pencil on paper manual responses. Each design receives from 0 to 2 points representing accuracy and location. Thus, scores range from 0 to 12. There are three learning trials. The outcome measure is the total number of points earned over the three trials.
The effect of rituximab on cognitive functions assessed by The California Verbal Learning Test-II | One year
  The California Verbal Learning Test-II (CVLT-II) begins with the examiner reading a list of 16 words. Patients listen to the list and report as many of the items as possible. After recall is recorded, the entire list is read again followed by a second attempt at recall. Altogether, there are five learning trials. The outcome measure is the total number of recalled items over the five trials.
The effect of rituximab on hand functions assessed by The Nine-Hole Peg Test | One year
  The Nine-Hole Peg Test (9-HPT) is a wood or plastic board with 9 holes (10 mm diameter, 15 mm depth) and a container. It is administered by asking the patient to take the pegs from a container, one by one, and place them into the holes on the board as quickly as possible. Participants must then remove the pegs from the holes, one by one, and replace them back into the container. The outcome measure is the time taken to complete the activity, recorded in seconds.

SECONDARY OUTCOMES:
The effect of rituximab on quality of life | One year
  Using MS-QLQ27 questionnaire, which contains 27 items covering physical, mental, and treatment-specific impairments as well as items relating to leisure, social, and work life issues. Scaling of items is a 5 point scale ranged from 1: "not at all impaired" to 5: "extremely impaired.
The effect of rituximab on EDSS | One year
  The Expanded Disability Status Scale (EDSS) is a tool used for quantifying disability in multiple sclerosis and monitoring changes in the level of disability over time. The scale ranges from 0 to 10 in 0.5 unit increments that represent higher levels of disability.

CONTACTS AND LOCATIONS:
Overall Officials: Maha Atef Zaki, MD Neurology, Study Chair — Department of Neurology, Faculty of Medicine, Cairo University; Amr Hassan Elsayed, MD Neurology, Study Chair — Department of Neurology, Faculty of Medicine, Cairo University
Locations (1):
- Kasr Alainy Multiple Sclerosis Unit (KAMSU), Cairo University hospitals., Giza, Giza Governorate, Egypt

IPD SHARING:
Plan to Share IPD: Yes
Analyzable IPD used in the results publication

REFERENCES:
- [Background] Carpinella I, Cattaneo D, Ferrarin M. Quantitative assessment of upper limb motor function in Multiple Sclerosis using an instrumented Action Research Arm Test. J Neuroeng Rehabil. 2014 Apr 18;11:67. doi: 10.1186/1743-0003-11-67. PMID 24745972
- [Background] Torgauten HM, Myhr KM, Wergeland S, Bo L, Aarseth JH, Torkildsen O. Safety and efficacy of rituximab as first- and second line treatment in multiple sclerosis - A cohort study. Mult Scler J Exp Transl Clin. 2021 Jan 31;7(1):2055217320973049. doi: 10.1177/2055217320973049. eCollection 2021 Jan-Mar. PMID 33796328
- [Background] Salehizadeh S, Saeedi R, Sahraian MA, Rezaei Aliabadi H, Hashemi SN, Eskandarieh S, Gheini MR, Shahmirzaei S, Owji M, Naser Moghadasi A. Effect of Rituximab on the cognitive impairment in patients with secondary progressive multiple sclerosis. Caspian J Intern Med. 2022 Summer;13(3):484-489. doi: 10.22088/cjim.13.3.484. PMID 35974939
- [Background] Naegelin Y, Naegelin P, von Felten S, Lorscheider J, Sonder J, Uitdehaag BMJ, Scotti B, Zecca C, Gobbi C, Kappos L, Derfuss T. Association of Rituximab Treatment With Disability Progression Among Patients With Secondary Progressive Multiple Sclerosis. JAMA Neurol. 2019 Mar 1;76(3):274-281. doi: 10.1001/jamaneurol.2018.4239. PMID 30615019
- [Background] Brochet B, Clavelou P, Defer G, De Seze J, Louapre C, Magnin E, Ruet A, Thomas-Anterion C, Vermersch P. Cognitive Impairment in Secondary Progressive Multiple Sclerosis: Effect of Disease Duration, Age, and Progressive Phenotype. Brain Sci. 2022 Jan 29;12(2):183. doi: 10.3390/brainsci12020183. PMID 35203948